CLINICAL TRIAL: NCT06005467
Title: The Effect of (v) Shaped Plate on Occlusion and Condylar Position Compared to Champy Technique in Fixation of Mandibular Angle Fracture (Randomized Clinical Trial)
Brief Title: V Shaped Plate Vs Champy Technique in Mandibular Angle Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Tohamy Abdelsattar Mohammed, Master's degree candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9793
Record Dates: First submitted 2023-07-06; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Fractures, Bone
Keywords: champy; angle fracture
MeSH Terms: conditions — Fractures, Bone | interventions — Open Fracture Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V shaped plate (Experimental): its a new plate that have been used in fixation of fractures in various areas of the mandible,V shaped plate was used in the treatment of three angle fracture cases which provided the advantage of including both lines of osteosynthesis which are the superior border and the lateral surface of the external oblique ridge using one plate.
  Interventions: Procedure: Open reduction and internal fixation of mandibular angle fracture using V shaped plate
- champy technique (Active Comparator): champy technique is one of the standard methods that are used in fixation of mandibular angle fractures by applying a mini-plate in the superior border of the external oblique ridge.
  Interventions: Procedure: Open reduction and internal fixation of mandibular angle fracture using V shaped plate

INTERVENTIONS:
Procedure: Open reduction and internal fixation of mandibular angle fracture using V shaped plate — its a new plate that have been used in fixation of fractures in various areas of the mandible,V shaped plate was used in the treatment of three angle fracture cases which provided the advantage of including both lines of osteosynthesis which are the superior border and the lateral surface of the external oblique ridge using one plate.

SUMMARY:
assessing fixation of mandibular angle fracture using two different mini plates, the standard champy technique and the new V shaped plate with comparing occlusion and condylar position between the two plates.

DETAILED DESCRIPTION:
The mandible is one of the most frequent bones of the face that is susceptible to fractures because its prominent position, as it comes in the second place after nasal fractures . Mostly, such fractures are a result of trauma caused by vehicle accidents, physical altercations, industrial accidents, falls, and contact sports, males usually suffer from mandibular fractures more than females.

The angle of the mandible is the most frequent area of the mandible to be fractured after the body, the reasons behind that is the presence of a third molar especially if it was impacted one which weakens the region even more, another reason is the existence of a very thin cross sectional area compared to the anterior parts of the mandible. Most common causes of mandibular angle fractures are motor vehicle collisions and assaults or altercations.

Therefore, the aim of this study is to evaluate a novel method which is using a (v) shaped plate in fixation of mandibular angle fracture, The new (v) shaped plate have provided easy reduction and stabilized fixation along both sides of the fracture, as it has two arms that can be easily adjusted over the angle of the mandible covering both lines of osteosynthesis along the superior border and lateral surface of the external oblique ridge using a single plate.

Although champy technique has been proven to be successful way for treating angle fractures with low complication rates it covers only one line of osteosynthesis which is the superior border of external oblique ridge unlike the (v) shaped plate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unilateral angle fracture.
2. Patients free from any systemic diseases that affect bone healing.
3. No sex predilection.
4. Age 18-50

Exclusion criteria:

1. Comminuted angle fractures.
2. Infected angle fracture.
3. Bilateral angle fracture.
4. Patients with any systemic diseases that affect bone healing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
proper occlusion | 1 week- 3 months and 6 months
  It's Clinically assessed outcome. Follow up will be carried out immediate post-operative (after1 week), 3months and after 6 months for general clinical assessment of the patient including proper occlusion.

SECONDARY OUTCOMES:
condylar position | 6 months
  C.T scan will be taken post operatively after periods of 1week and 6 months to measure condylar position by specialized (software mimics) C.T superimposition.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhagat MJA, Durairaj D, Naganathan V, Nathiya B, Kumar GS, Mariam S. Application of Anatomically Designed 2-Dimensional V Plate in Management of Mandible Fracture: A Pilot Study. J Maxillofac Oral Surg. 2022 Dec;21(4):1363-1368. doi: 10.1007/s12663-021-01558-5. Epub 2021 Apr 23. PMID 36896057
- [Background] Lee JH. Treatment of Mandibular Angle Fractures. Arch Craniofac Surg. 2017 Jun;18(2):73-75. doi: 10.7181/acfs.2017.18.2.73. Epub 2017 Jun 26. PMID 28913310